CLINICAL TRIAL: NCT03538483
Title: Erector Spinae Plane Block Versus Serratus Plane Block on Postoperative Opioid Consumption for Modified Radical Mastectomy and Axillary Lymph Node Dissection
Brief Title: Erector Spinae Plane Block Versus Serratus Plane Block for Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUTFANESTHESIA
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Pain; Breast Cancer
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided serratus plane block (Active Comparator): Ultrasound Guided Serratus Plane Block 30 ml %0.25 Bupivacaine
  Interventions: Drug: Bupivacaine Hcl 0.25% Inj
- ultrasound guided erector spinae plane block (Active Comparator): Ultrasound Guided Erector Spinae Plane Block 20 ml %0.25 Bupivacaine
  Interventions: Drug: Bupivacaine HCl Inj 0.25%

INTERVENTIONS:
Drug: Bupivacaine Hcl 0.25% Inj — 30 ml %0,25 bupivacaine
  Arms: ultrasound guided serratus plane block
Drug: Bupivacaine HCl Inj 0.25% — 20 ml %0,25 bupivacaine
  Arms: ultrasound guided erector spinae plane block

SUMMARY:
Serratus plane block (SPB) was first described in 2013 by Blanco and designed to primarily block the thoracic intercostal nerves. And this block provides sufficient analgesia lateral anterior and posterior part of thoracic wall.Erector Spinae Plane Block (ESPB) is a newly described and effective interfascial plane block for thoracic and abdominal surgery. It was first described by Forero et al. in 2016, effectiveness being reported in four cases. The aim of this study is to compare Serratus plane block and erector spinae plane block on postoperative pain in patients undergoing modified radical mastectomy and axillary lymph node dissection

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients
* undergoing breast cancer surgery
* 18-65 years

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications
* emergency cases
* coagulopathy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | First 24 hours
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | postoperative first24 hours
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain) at first hour postoperatively
Block Performing Time | First hour
  The block time was defined as the period between the insertion of the needle and termination of local anesthetic administration

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No